CLINICAL TRIAL: NCT01928810
Title: The Influence of Physical Activity (Prior to In-vivo Exposure) on the Effect of Cognitive Behavioural Therapy in Patients With Panic Disorder and Agoraphobia
Brief Title: Physical Activity and Cognitive Behavioural Therapy in Panic Disorder and Agoraphobia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Ströhle, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201015
Record Dates: First submitted 2013-07-26; First posted 2013-08-27 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Panic Disorder; Agoraphobia
Keywords: Panic Disorder; Agoraphobia; Physical Activity
MeSH Terms: conditions — Panic Disorder; Agoraphobia; Motor Activity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 70% VO2max (Experimental): Cognitive Behavioural Therapy (CBT)
  + aerobic exercise (30 minutes, 70% VO2max) prior to 5 in-vivo exposure sessions
  Interventions: Behavioral: Cognitive Behavioural Therapy
- 30% VO2max (Active Comparator): Cognitive Behavioural Therapy (CBT)
  + placebo exercise (30 minutes, 30% VO2max) prior to 5 in-vivo exposure sessions
  Interventions: Behavioral: Cognitive Behavioural Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy — 12 sessions of CBT including psychoeducation, interoceptive exposure and in-vivo exposure
  Other Names: CBT

SUMMARY:
Physical activity (treadmill) prior to in-vivo exposure supports the effect of cognitive behavioural therapy in patients with panic disorder and agoraphobia.

DETAILED DESCRIPTION:
Patients receive a 12-session manualized cognitive behavioural therapy, implemented over 7 weeks and followed by two booster sessions. Five sessions consist of in-vivo exposures. Prior to these sessions patients undergo a training of physical activity. Half of the patients complete training on a treadmill at 70% of their maximal oxygen uptake while the other half complete training at 30%.

ELIGIBILITY:
Inclusion Criteria:

* Subject familiarized with experimental procedure and had given written informed consent
* Diagnosis of panic disorder with agoraphobia according to Diagnostic and Statistical Manual of Mental Disorders (DSM-IV)
* Score >= 18 in Hamilton Rating Scale for Anxiety
* Score >= 4 in Clinical Global Index
* Reachability of patient for treatment and follow-up

Exclusion Criteria:

* DSM-IV Axis I diagnoses of any psychotic disorder, bipolar disorder, current alcohol or drug dependence and Axis II borderline personality disorder
* Change in pharmacological treatment in the last 4 weeks
* Acute suicidality
* Medical contraindications for mild to moderate exercise training or exposure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Anxiety (CIPS 1995) | Change from Baseline to 31 weeks (follow-up)
  Global interviewer rated measure for anxiety and severity indicator of an anxiety disorder
Mobility Inventory (Chambless 1984) | Change from Baseline to 31 weeks (follow-up)
  A 27-item inventory for the measurement of self-reported agoraphobic avoidance behavior

SECONDARY OUTCOMES:
Clinical Global Index (CIPS 1995) | Baseline, 3 weeks, 7 weeks, 31 weeks (follow up)
Beck Depression Inventory (CIPS 1995) | Baseline, 3 weeks, 7 weeks, 31 weeks (follow up)
Anxiety Sensitivity Index (Taylor 1998) | Baseline, every second session, 3 weeks, 7 weeks, 31 weeks (follow up)
Body Sensations Questionnaire (Chambless 1984) | Baseline, 3 weeks, 7 weeks, 31 weeks (follow up)
Agoraphobic Cognitions Questionaire (Chambless 1984) | Baseline, 3 weeks, 7 weeks, 31 weeks (follow up)
Panic and Agoraphobia Scale | Change from baseline to 31 weeks (follow-up)
  Severity scale for panic disorder

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Bischoff, Dipl.-Psych., Principal Investigator — Charite

REFERENCES:
- See also: Related Info — http://www.angstambulanz-charite.de/